CLINICAL TRIAL: NCT04701190
Title: Comparison of Different Noradrenaline Protocols to Prevent Post Spinal Hypotension During Elective Caesarean Delivery: A Randomised, Double-blind Clinical Trial
Brief Title: Different Noradrenaline Protocols in Post Spinal Hypotension in CS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Menekse Ozcelik, Associate Professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Hypotension; Cesarean Section; Anesthesia, Spinal
Keywords: Apgar Score; Pregnancy; Blood Pressure; Heart Rate; adult; female; Hypotension; Noradrenaline; Cesarean Section; Anesthesia, Spinal
MeSH Terms: conditions — Hypotension | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The hypotension will be recognized by the participants due to feeling unwell of theirselves. However they will not have any information about the dosage of the study drug. So they will be blinded to the study group which they will be included by the investigator of the study.
  The investigator will collect the data coming from the monitors, patients and the newborn. Therefore, the investigator will not be aware of the intervention about the dosing of noradrenaline made by the anesthesiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Noradrenaline 0.05/10 (Active Comparator): Study drug will be prepared as follows:4 milligram noradrenaline will be administered into 100 milliliter 5% dextrose solution.
  The basal blood pressure of the parturient will be recorded as an arithmetic sum of the sequential three measurements of noninvasive blood pressure.
  Maternal hypotension and severe hypotension will be described as a decrease of noninvasive systolic blood pressure according to basal systolic blood pressure by 20% and 40%, respectively.
  If the heart rate of parturient will be under 60 beat/minute, this will be recorded as maternal bradycardia.
  The noradrenaline bolus dosage of 10 microgram will be administered to the patient at the same time of obtaining cerebrospinal fluid running freely. After the end of the injection of heavy marcaine 0.5% to the subarachnoid space, the infusion of noradrenaline with a 0.05 microgram/kg/minute dosage will be started.
  Noradrenaline will be continued until 5 minutes after delivery of fetus.
  Interventions: Drug: Noradrenalin 10 microgram bolus; Drug: Noradrenaline 0.05 microgram/kg/minute infusion; Procedure: Spinal anesthesia
- Noradrenaline 0.075/5 (Active Comparator): Study drug will be prepared as follows:4 milligram noradrenaline will be administered into 100 milliliter 5% dextrose solution.
  The basal blood pressure of the parturient will be recorded as an arithmetic sum of the sequential three measurements of noninvasive blood pressure.
  Maternal hypotension and severe hypotension will be described as a decrease of noninvasive systolic blood pressure according to basal systolic blood pressure by 20% and 40%, respectively.
  If the heart rate of parturient will be under 60 beat/minute, this will be recorded as maternal bradycardia.
  The noradrenaline bolus dosage of 5 microgram will be administered to the patient at the same time of obtaining cerebrospinal fluid running freely. After the end of the injection of heavy marcaine 0.5% to the subarachnoid space, the infusion of noradrenaline with a 0.075 microgram/kg/minute dosage will be started.
  Noradrenaline will be continued until 5 minutes after delivery of fetus.
  Interventions: Drug: Noradrenaline 5 microgram bolus; Drug: Infusion dosage: 0.075 microgram/kg/minute infusion; Procedure: Spinal anesthesia
- Noradrenaline 0.1/0 (Active Comparator): Study drug will be prepared as follows:4 milligram noradrenaline will be administered into 100 milliliter 5% dextrose solution.
  The basal blood pressure of the parturient will be recorded as an arithmetic sum of the sequential three measurements of noninvasive blood pressure.
  Maternal hypotension and severe hypotension will be described as a decrease of noninvasive systolic blood pressure according to basal systolic blood pressure by 20% and 40%, respectively.
  If the heart rate of parturient will be under 60 beat/minute, this will be recorded as maternal bradycardia.
  After the end of the injection of heavy marcaine 0.5% to the subarachnoid space, the infusion of noradrenaline with a 0.1 microgram/kg/minute without bolus dosage will be started.
  Noradrenaline will be continued until 5 minutes after delivery of fetus.
  Interventions: Drug: Noradrenaline 0.1 microgram/kg/minute infusion; Procedure: Spinal anesthesia

INTERVENTIONS:
Drug: Noradrenalin 10 microgram bolus — The noradrenaline bolus dosage of 10 microgram will be administered to the patient at the same time of obtaining cerebrospinal fluid running freely.
  Other Names: NA 10B
  Arms: Noradrenaline 0.05/10
Drug: Noradrenaline 5 microgram bolus — The noradrenaline bolus dosage of 5 microgram will be administered to the patient at the same time of obtaining cerebrospinal fluid running freely.
  Other Names: NA 5B
  Arms: Noradrenaline 0.075/5
Drug: Noradrenaline 0.1 microgram/kg/minute infusion — Infusion dosage: 0.1 microgram/kg/minute After the end of the injection of heavy marcaine 0.5% to the subarachnoid space, the infusion of noradrenaline with a 0.1 microgram/kg/minute dosage will be started.
  Noradrenaline will be continued until 5 minutes after delivery of fetus.
  Other Names: NA 0.1I
  Arms: Noradrenaline 0.1/0
Drug: Noradrenaline 0.05 microgram/kg/minute infusion — Infusion dosage: 0.05 microgram/kg/minute After the end of the injection of heavy marcaine 0.5% to the subarachnoid space, the infusion of noradrenaline with a 0.05 microgram/kg/minute dosage will be started.
  Noradrenaline will be continued until 5 minutes after delivery of fetus.
  Other Names: NA 0.05I
  Arms: Noradrenaline 0.05/10
Drug: Infusion dosage: 0.075 microgram/kg/minute infusion — nfusion dosage: 0.075 microgram/kg/minute After the end of the injection of heavy marcaine 0.5% to the subarachnoid space, the infusion of noradrenaline with a 0.075 microgram/kg/minute dosage will be started.
  Noradrenaline will be continued until 5 minutes after delivery of fetus.
  Other Names: NA 0.075I
  Arms: Noradrenaline 0.075/5
Procedure: Spinal anesthesia — Spinal anesthesia using 0.5% 10 milligram heavy bupivacaine plus 12.5 microgram fentanyl

SUMMARY:
The incidence of hypotension after spinal anesthesia is approximately 60% in parturients undergoing cesarean section. As a consequence of hypotension, nausea-vomiting, dyspnea and neurological deterioration in patients and low Apgar scores in newborns may occur. Therefore, there is an increasing interest to prevent maternal post spinal hypotension by using several drugs including noradrenaline given in different protocols to the patients undergoing spinal anesthesia for cesarean section. However, there is no conclusive answer to the question of which dosage is the best to prevent the maternal post spinal hypotension in literature.

In this prospective randomized study, we aimed to compare different noradrenaline protocols for preventing maternal post spinal hypotension during elective cesarean delivery.

DETAILED DESCRIPTION:
One of the most important and frequent adverse effects of spinal anesthesia is post procedure hypotension. The emerging hypotension does not affect only the pregnant, it also does harm to the newborn. Therefore, an anesthesiologist should avoid and take precautions to prevent maternal post spinal hypotension. There is a growing body of evidence about noradrenalin application in the management of hemodynamic optimization of patients undergoing cesarean section with spinal anesthesia. However, there is no conclusive decision about the dosage and application protocol of noradrenaline in this patient population. In a study comparing the incidence of post spinal maternal hypotension given noradrenaline versus phenylephrine, the authors reported that both of drugs effectively controlled maternal blood pressure. The incidence of maternal hypotension was 30% and 32% (p= 0.8) in noradrenaline and phenylephrine study arms, respectively. Therefore, one can speculate that the incidence of maternal post spinal hypotension remains high even in patients receiving noradrenaline or phenylephrine. In the noradrenaline arm, only noradrenaline infusion with a dosage of 0.05 microgram/kg/minute without any bolus was applied to the patients. In another study, the effects of different noradrenaline infusion dosages with 5 microgram bolus dosage on maternal post spinal hypotension were investigated. The frequencies of maternal hypotension were 42.1%, 24.7% and 26% in patients receiving 0.025, 0.05 and 0.075 microgram/kg/minute with a bolus 5 microgram noradrenaline, respectively. As a conclusion of this study, addition of a bolus dose of 5 microgram noradrenaline may lower the incidence of post spinal hypotension. However, as in the previous study, approximately one fourth of patients still may have a post spinal hypotension episode. Regarding these results, the present study is planned to answer the question of which approach including increasing infusion or bolus dosage of noradrenaline is superior to ameliorate the incidence of hypotension in this population.

In conclusion, the aim of this study is to compare three different noradrenaline protocols including different bolus and infusion dosages to decrease the rate of hypotension in patients undergoing cesarean section with spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA 2
* 38 +4 gestational age parturient

Exclusion Criteria:

* ASA 3-6
* Parturients with any kind of contraindication to spinal anesthesia
* Hypertensive parturients (basal systolic blood pressure above 140 mmHg)
* Parturients having basal systolic blood pressure below 100 mmHg
* Parturients having peripartum hemorrhage
* Parturients having body mass index above 40
* Parturients with a known allergic reaction to one of the study drugs
* Parturients not willing to be included into the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Parturient
Enrollment: 180 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of maternal post spinal hypotension | Between the application time of spinal anesthesia and 5th minute after delivery
  The primary outcome of this study is to compare the incidences of maternal post spinal hypotension in patients administered three different noradrenaline protocols.
Incidence of maternal post spinal severe hypotension | Between the application time of spinal anesthesia and 5th minute after delivery
  The other primary outcome of this study is to compare the incidences of maternal post spinal severe hypotension in patients administered three different noradrenaline protocols.

SECONDARY OUTCOMES:
The incidence of post delivery maternal hypotension | Between 5th minute after delivery and the end of surgery
  The secondary outcome of this study is to compare the incidences of maternal post delivery hypotension in patients administered three different noradrenaline protocols.
The incidence of post delivery maternal severe hypotension | Between 5 minute of delivery and the end of surgery
  The other secondary outcome of this study is to compare the incidences of maternal post delivery severe hypotension in patients administered three different noradrenaline protocols.
The incidence of intervention applied by an anesthesiologist | Between the start of patient monitoring and the end of surgery
  The other secondary outcome is to determine and to compare the frequency of intervention applied by the anesthesiologist to stabilize the patients hemodynamic status.This interventions include changing the noradrenaline infusion status, administering atropine and ephedrine, according to the patients hemodynamic data.

CONTACTS AND LOCATIONS:
Overall Officials: Menekse Ozcelik, M.D, Principal Investigator — Associate Professor
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vallejo MC, Attaallah AF, Elzamzamy OM, Cifarelli DT, Phelps AL, Hobbs GR, Shapiro RE, Ranganathan P. An open-label randomized controlled clinical trial for comparison of continuous phenylephrine versus norepinephrine infusion in prevention of spinal hypotension during cesarean delivery. Int J Obstet Anesth. 2017 Feb;29:18-25. doi: 10.1016/j.ijoa.2016.08.005. Epub 2016 Aug 28. PMID 27720613
- [Background] Hasanin AM, Amin SM, Agiza NA, Elsayed MK, Refaat S, Hussein HA, Rouk TI, Alrahmany M, Elsayad ME, Elshafaei KA, Refaie A. Norepinephrine Infusion for Preventing Postspinal Anesthesia Hypotension during Cesarean Delivery: A Randomized Dose-finding Trial. Anesthesiology. 2019 Jan;130(1):55-62. doi: 10.1097/ALN.0000000000002483. PMID 30335625
- [Background] Hasanin A, Amin S, Refaat S, Habib S, Zayed M, Abdelwahab Y, Elsayad M, Mostafa M, Raafat H, Elshall A, Fatah SAE. Norepinephrine versus phenylephrine infusion for prophylaxis against post-spinal anaesthesia hypotension during elective caesarean delivery: A randomised controlled trial. Anaesth Crit Care Pain Med. 2019 Dec;38(6):601-607. doi: 10.1016/j.accpm.2019.03.005. Epub 2019 Mar 30. PMID 30935897
- [Derived] Baytas V, Karadag Erkoc S, Ozcelik M, Gokmen D, Bermede AO, Selvi Can O, Uysalel A. A Randomized, Double-Blind, Graded Dose-Response Study of Norepinephrine Administration for Prevention of Post-Spinal Hypotension during Elective Cesarean Delivery. J Clin Med. 2023 Oct 10;12(20):6437. doi: 10.3390/jcm12206437. PMID 37892573